CLINICAL TRIAL: NCT07199582
Title: Association Between Obesity and Gastroesophageal Reflux Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dina Adolf Habib Khela, residant doctor at Assiut university hospital, Assiut University
Other Study IDs: GERD and Obesity
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Gastro Esophageal Reflux; Obesity (Disorder)
MeSH Terms: conditions — Gastroesophageal Reflux; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: obese patients
- Group B: non obese patients

SUMMARY:
Gastroesophageal reflux disease (GERD) is a chronic disorder marked by heartburn and regurgitation, resulting from the reflux of gastric acid or bile into the esophagus. Chronic acid exposure leads to mucosal inflammation, erosive esophagitis, and Barrett's esophagus, conditions that increase the risk of esophageal adenocarcinoma (Badreddine RJ et al., 2010; Fass R, 2022). Obesity, defined by the World Health Organization as a body mass index (BMI) ≥30 kg/m², is recognized as a major global public health issue due to its rapidly rising prevalence and strong association with chronic disease. It is not only a cause of metabolic disorders but also a driver of systemic health complications (WHO, 2024). Obesity is linked with type 2 diabetes, cardiovascular disease, hypertension, non-alcoholic fatty liver disease, certain cancers, and sleep apnea.

Additionally, it negatively impacts psychological well-being, contributing to depression, low self-esteem, and social stigma (CDC, 2024). Evidence suggests a strong link between obesity and GERD. Studies demonstrate that obese individuals exhibit higher intra-gastric pressure, delayed esophageal transit, increased esophageal acid exposure, and a greater prevalence of defective lower esophageal sphincter function. These pathophysiological mechanisms contribute significantly to GERD development and its complications (de Vries DR et al., 2008; Cote-Daigneault J et al., 2014; Anggiansah R et al., 2013; Ayazi S et al., 2009). The rationale for this study is to explore the relationship between obesity and GERD, given the rising prevalence of obesity and its implications for gastrointestinal health. Diagnosis of GERD is primarily clinical, based on symptoms such as heartburn and regurgitation. A trial of proton pump inhibitors for 4-8 weeks is recommended in patients without alarm features. Endoscopy is indicated for those with alarm signs or refractory disease, while pH monitoring is the gold standard in uncertain cases. Manometry is reserved for pre-surgical evaluation (Katz PO et al., 2022).To study the relationship between Obesity and GERD, given the rising prevalence of obesity and its potential impact on gastrointestinal health.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old. Obese patients (BMI ≥30 Kg/m2).

Exclusion Criteria:

* · Eosinophilic esophagitis.

  * Achalasia.
  * Esophageal cancer. Stomach cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: obese patients aged >18 years with BMI>30 kg
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
prevalence of obesity | Baseline
  the prevalence of obesity among GERD patients